CLINICAL TRIAL: NCT01029730
Title: Phase II Trial of Bendamustine, Bortezomib, and Rituximab in Patients With Previously Untreated Low Grade Lymphoma
Brief Title: Trial of Bendamustine, Bortezomib, and Rituximab in Patients With Previously Untreated Low Grade Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LYM 66
Record Dates: First submitted 2009-12-08; First posted 2009-12-10 (Estimated); Results first posted 2015-12-28 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: Low grade lymphoma; Previously untreated lymphoma; Lymphoma first line; bendamustine; Treanda; bortezomib; Velcade; rituximab; Rituxan
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride; Bortezomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine/Bortezomib/Rituximab (Experimental): Treatment for all patients will be given in cycles of 28 days (4 weeks). All patients will receive treatment with bendamustine, bortezomib, and rituximab for a maximum of 6 cycles. Rituximab should be administered first.
  Interventions: Drug: Bendamustine; Drug: Bortezomib; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine — Bendamustine: 90 mg/m2 Days 1 and 2 of 6, 28-day cycles
  Other Names: TREANDA®
Drug: Bortezomib — Bortezomib: 1.6 mg/m2 given IV on Day 1, Day 8, and Day 15 of 6, 28-day cycles
  Other Names: VELCADE®
Drug: Rituximab — Rituximab, Cycle 1: 375 mg/m2 given IV on Day 1, Day 8, and Day 15 Rituximab, Cycles 2-6: 375 mg/m2 given IV on Day 1
  Other Names: Rituxan®

SUMMARY:
The goal of this multi-center Phase II study is to add bortezomib to the highly active regimen of bendamustine and rituximab. In this study, bortezomib will be administered on a weekly schedule (Days 1, 8, 15) and will be added to bendamustine/rituximab given in 4-week cycles. This combination uses the standard bendamustine dosing schedule, and is more convenient than the 5-week regimen of these 3 drugs currently being studied.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed indolent lymphoma by the World Health Organization (WHO) classification. The biopsy must fulfill one of the following criteria:

   * Follicular lymphoma, grade 1 or 2
   * Marginal zone lymphoma
   * Small lymphocytic lymphoma (circulating lymphocyte count must be <5,000)
   * Lymphoplasmacytic lymphoma
2. At least one of the following criteria must be met:

   * Presence of any symptoms related to lymphoma. These can include classic B-symptoms (fever [>38°C] of unclear etiology, night sweats, weight loss of greater than 10% within the prior 6 months) or other lymphoma-related symptoms (fatigue, pain, etc.).
   * Large tumor mass (bulky disease) characterized by lymphomas with a diameter of more than 3 cm in three or more regions or by a lymphoma with a diameter >7 cm in one region
   * Presence of lymphoma-related complications, including narrowing of ureters or bile ducts, tumor-related compression of a vital organ, lymphoma-induced pain, cytopenias related to lymphoma/leukemia, splenomegaly, pleural effusions, or ascites
   * Hyperviscosity syndrome due to monoclonal gammopathy
3. The lymph node biopsy or other lymphoma pathology specimen has CD20+ B-cells.
4. Ann-Arbor Stage 2 (non-contiguous), 3, or 4 disease.
5. No previous systemic treatment for lymphoma. Patients may have had a single course of radiation therapy to a limited field (i.e., not exceeding two adjacent lymph node regions).
6. The patient has bidimensionally measurable disease with at least 1 lesion measuring ≥2.0 cm in a single dimension, and the field was not previously radiated.
7. An Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
8. Adequate hematologic function ≤7 days prior to start of study treatment:

   * Hemoglobin ≥10.0 g/dl
   * Absolute neutrophil count (ANC) ≥1000/µL
   * Platelet count ≥75,000/µL. If low counts are attributable to bone marrow infiltration or hypersplenism due to lymphoma, ANC must be ≥750/µL and platelets ≥50,000/µL.
9. Calculated or measured creatinine clearance ≥30 mL/min ≤7 days of study enrollment (using Cockcroft-Gault method).
10. Adequate hepatic function (≤2.5 x upper limit of normal [ULN] for alanine aminotransferase [ALT], aspartate aminotransferase [AST], and alkaline phosphatase and total bilirubin within normal limits).
11. Patients must be ≥18 years of age.
12. Women of childbearing potential must agree to use a medically acceptable method of birth control (e.g., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and for 12 months after their last dose of rituximab. Men must use an acceptable method/form of contraception for the duration of treatment and for 3 months after the end of treatment.
13. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.

Exclusion Criteria:

1. The patient has chronic lymphocytic leukemia.
2. The patient has transformed lymphoma.
3. History of, or clinically apparent, central nervous system (CNS) lymphoma or leptomeningeal lymphoma.
4. The patient has received corticosteroids for treatment of lymphoma. Chronic, low-dose corticosteroids (e.g., prednisone ≤20 mg/day) are allowed for treatment uses other than lymphoma or complications of lymphoma.
5. Peripheral neuropathy ≥ CTCAE v3.0 grade 2, ≤14 days of study enrollment.
6. Myocardial infarction ≤6 months prior to study enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, ECG abnormalities at screening must be documented as not medically relevant.
7. History of solid organ transplantation, or post-transplant lymphoproliferative disorder.
8. Patients with known history of hepatitis B or hepatitis C infection. Hepatitis B surface antigen must be tested.
9. The patient has known human immunodeficiency virus (HIV) infection.
10. Active, clinically serious infection > grade 2. Patients may be eligible upon resolution of the infection.
11. Female patient is pregnant or breast-feeding. Confirmation that female patients of childbearing potential are not pregnant must be established by a negative serum pregnancy test ≤7 days prior to the start of treatment.
12. Known hypersensitivity to bendamustine, bortezomib, boron, mannitol, or rituximab.
13. Concomitant active malignancy requiring therapy.
14. Diagnosis or treatment for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
15. Treatment with other investigational agents ≤14 days prior to study enrollment.
16. Any other disease(s), psychiatric condition, metabolic dysfunction, or findings from a physical examination or clinical laboratory test result that would cause reasonable suspicion of a disease or condition, that contraindicates the use of study drugs, that may increase the risk associated with study participation, that may affect the interpretation of the results, or that would make the patient inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-03; Primary Completion 2014-10 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian W. Flinn, MD, PhD, Study Chair — SCRI Development Innovations, LLC
Locations (20):
- United States (20):
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Hematology Oncology of the North Shore, Skokie, Illinois
  - Providence Medical Group, Terre Haute, Indiana
  - Baptist Hospital East, Louisville, Kentucky
  - Hematology Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Schiffler Cancer Center, Wheeling, West Virginia

RESULTS

PARTICIPANT FLOW:
Period: Combination Therapy
Arm/Group | Bendamustine/Bortezomib/Rituximab
Started | 55
Completed | 39 (Patients remained on-study until completing 6 cycles or coming off-treatment for any other reason)
Not Completed | 16
Period: Maintenance Therapy
Arm/Group | Bendamustine/Bortezomib/Rituximab
Started | 37 (Two patients complete study treatment but declined subsequent maintenance therapy)
Completed | 14
Not Completed | 23

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Arm/Group | Bendamustine/Bortezomib/Rituximab
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 64 [30 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Percentage of patients experiencing a complete response (CR) per RECIST. CR = disappearance of all target lesions.
Time Frame: 18 months
Population: All evaluable patients
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Bendamustine/Bortezomib/Rituximab
Number analyzed (Participants) | 51
percentage of evaluable participants | 65

2. Secondary Outcome: Overall Response Rate
Description: The Percentage of Patients Who Experience an Objective Benefit From Treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: At 3 and 6 months during treatment, then 6 months post-treatment.
Population: All patients evaluable for response.
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Bendamustine/Bortezomib/Rituximab
Number analyzed (Participants) | 51
percentage of evaluable participants | 94

3. Secondary Outcome: Median Progression-free Survival
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: at 3 and 6 months, then every 3 months post-treatment for 1 year and every 6 months thereafter until disease progression; projected 2 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine/Bortezomib/Rituximab
Number analyzed (Participants) | 55
months | NA [NA to NA] — Median PFS was not reached

4. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety.
Description: Toxicity grades will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0. Includes adverse events occurring in >1 patient
Time Frame: Days 1,8, and 15 of each 28-day cycle for 6 months, then every 3 months for a year, projected 2 years.
Population: All patients
Measure: Number; unit: participants
Arm/Group | Bendamustine/Bortezomib/Rituximab
Number analyzed (Participants) | 55
participants
  Leukopenia | 16
  Neutropenia | 16
  Lymphopenia | 9
  Thrombocytopenia | 4
  Anemia | 3
  Peripheral Neuropathy | 5
  Diarrhea | 4
  Fatigue | 4
  Nausea/Vomiting | 3
  Cough | 2
  Rash | 2
  Syncope | 2
  Hypocalcemia/Hyponatremia | 2

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Bendamustine/Bortezomib/Rituximab
Serious Adverse Events (participants affected / at risk) | 11/55
Other Adverse Events (participants affected / at risk) | 54/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine/Bortezomib/Rituximab (N=55)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac disorders - other, left ventricular diastolic dysfunction (Cardiac disorders) | 1
Cardiac disorders - Other, tachycardia (Cardiac disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Fever (General disorders) | 1
Gastrointestinal disorders - Other, bowel perforation (Gastrointestinal disorders) | 1
Hepatitis viral (Infections and infestations) | 1
Infections and infestations - Other, Perisigmoid abscess (Infections and infestations) | 1
Infections and infestations - Other, Varicella (Infections and infestations) | 1
Infusion Related Reaction (General disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Skin Infection (Infections and infestations) | 1
Tremor (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine/Bortezomib/Rituximab (N=55)
Fatigue (General disorders) | 48
Nausea (Gastrointestinal disorders) | 39
Platelet Count Decreased (Investigations) | 34
White Blood Cell Decreased (Investigations) | 30
Constipation (Gastrointestinal disorders) | 29
Peripheral Sensory Neuropathy (Nervous system disorders) | 29
Anemia (Blood and lymphatic system disorders) | 25
Diarrhea (Gastrointestinal disorders) | 25
Neutrophil Count Decreased (Investigations) | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 23
Hyperglycemia (Metabolism and nutrition disorders) | 21
Vomiting (Gastrointestinal disorders) | 18
Rash (Skin and subcutaneous tissue disorders) | 18
Edema (General disorders) | 15
Insomnia (Psychiatric disorders) | 15
Anorexia (Metabolism and nutrition disorders) | 14
Dizziness (Nervous system disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Lymphocyte Count Decreased (Investigations) | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 12
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 12
Fever (General disorders) | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Chills (General disorders) | 10
Headache (Nervous system disorders) | 10
Tinnitus (Ear and labyrinth disorders) | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 9
Mucositis (Gastrointestinal disorders) | 8
Pain (General disorders) | 8
Dysgeusia (Nervous system disorders) | 8
Infections And Infestations - Other, Herpes Zoster (Infections and infestations) | 8
Abdominal Pain (Gastrointestinal disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 7
Allergic Reaction (Immune system disorders) | 6
Infections And Infestations - Other, Unspecified (Infections and infestations) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 6
Anxiety (Psychiatric disorders) | 6
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 6
Alanine Aminotransferase Increased (Investigations) | 6
Flatulence (Gastrointestinal disorders) | 5
Alkaline Phosphatase Increased (Investigations) | 5
Aspartate Aminotransferase Increased (Investigations) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Depression (Psychiatric disorders) | 5
Hypertension (Vascular disorders) | 5
Investigations - Other, Ldh Increased (Investigations) | 5
Abdominal Distension (Gastrointestinal disorders) | 4
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 4
Upper Respiratory Infection (Infections and infestations) | 4
Weight Loss (Investigations) | 4
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4
Investigations - Other, Creatinine Decreased (Investigations) | 4
Investigations - Other, Blood Protein Decreased (Investigations) | 4
Dry Mouth (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 3
Flu Like Symptoms (General disorders) | 3
Bronchial Infection (Infections and infestations) | 3
Infections And Infestations - Other, Oral Infection (Infections and infestations) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 3
Urinary Frequency (Renal and urinary disorders) | 3
Pelvic Pain (Reproductive system and breast disorders) | 3
Respiratory, Thoracic And Mediastinal Disorders - Other, Runny Nose (Respiratory, thoracic and mediastinal disorders) | 3
Hot Flashes (Vascular disorders) | 3
Investigations - Other, Blood Bicarbonate Increased (Investigations) | 3
Injection Site Reaction (General disorders) | 3
Investigations - Other, Ldh Increased (Investigations) | 3
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites